CLINICAL TRIAL: NCT04771806
Title: Serial Advanced Magnetic Resonance Imaging (MRI) for Guidance of Personalized Adaptive Radiotherapy for High Grade Glioma
Brief Title: Serial Advanced Magnetic Resonance Imaging Scan for Guidance of Personalized Adaptive Radiotherapy for High Grade Glioma
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA17-0844; NCI-2020-08129 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA17-0844 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-12-20; First posted 2021-02-25 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Malignant Glioma
MeSH Terms: conditions — Glioma | interventions — Magnetic Resonance Spectroscopy; Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Observational (MRI): Patients undergo MRI with and without contrast immediately before radiotherapy (for radiation planning) and at mid treatment (week 3). Patients also undergo MRI without contrast on weeks 1, 2, 4, 5, and 6 of radiotherapy. Patients may also undergo neurocognitive function testing over 70 minutes before treatment, at the end of each week of treatment, and at 3 and 6 months after completion of treatment.
  Interventions: Procedure: Magnetic Resonance Imaging; Other: Neurocognitive Assessment; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Other: Neurocognitive Assessment — Undergo neurocognitive testing
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This study examines whether repeated magnetic resonance imaging (MRI)s scan helps identify changes in the tumor during radiation and chemotherapy treatment in patients with high grade glioma. Additional MRIs scan may help researchers to see changes in the status of the disease. Seeing these changes may result in changes to the treatment plan.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the radiation dosimetric coverage of the surgical cavity and any residual tumor when the immediate post-operative MRI is used versus (vs.) newly acquired MRI prior to radiation therapy.

II. To evaluate the cumulative dosimetric differences for the target volume and normal structures between an adaptive radiotherapy approach based on serial MRI vs. the conventionally delivered radiotherapy plan using the target and normal structure volumes from the initial MRI simulation.

SECONDARY OBJECTIVES:

I. To report the incidence of tumor progression between surgery and radiation therapy and factors related to higher risk of tumor progression (e.g. Time interval between surgery and radiation, extent of surgery, molecular characteristics).

II. To evaluate the relationship between the delivered dosimetry and patterns of failure and changes in neurocognitive function.

III. To evaluate the relationship between voxel-wise quantitative changes on multiparametric MRI including apparent diffusion coefficient (ADC), fractional anisotropy (FA), relative cerebral blood volume (rCBV), fractional volume of the extravascular, extracellular space (ve) and Ktrans (transfer constant that characterizes the diffusive transport of low-molecular weight gadolinium across the capillary endothelium) with patterns of failure and changes in neurocognitive function.

IV. To determine if early post-operative progression is associated with worse overall survival.

V. To determine the difference in reported pseudoprogression at first follow-up after completing radiation when the baseline MRI is the immediate post-op MRI vs. newly acquired MRI prior to radiation therapy.

VI. To compare image co-registration accuracy between the radiation planning computed tomography (CT) images and MRI for the immediate post-op MRI vs. newly acquired MRI prior to radiation therapy.

VII. To evaluate the relationship between standard clinical neurocognitive function (NCF) and iPad based NCF (iNCF) test results.

OUTLINE:

Patients undergo MRI with and without contrast immediately before radiotherapy (for radiation planning) and at mid treatment (week 3). Patients also undergo MRI without contrast on weeks 1, 2, 4, 5, and 6 of radiotherapy. Patients may also undergo neurocognitive function testing over 70 minutes before treatment, at the end of each week of treatment, and at 3 and 6 months after completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients with histologic confirmation of high grade glioma
* Patients must be age >= 18 years
* Patients must sign informed consent indicating that they are aware of the investigational nature of this study in keeping with the policies of the hospital. The only acceptable consent form is the one attached at the end of this protocol, and has been approved and amended by the MD Anderson Cancer Center (MDACC) Institutional Review Board (IRB)
* Patients must have Karnofsky performance status (KPS) >= 60
* Patients must be able to obtain an MRI scan with gadolinium contrast
* Female patients of childbearing age must not be pregnant as determined with a serum beta human chorionic gonadotropin (HCG) no greater than 14 days prior to study registration, or breastfeeding. (The exclusion is made because gadolinium may be teratogenic in pregnancy). Female patients who consent to participate in the study will need to use contraceptive methods for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologic confirmation of high grade glioma
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Differences in the delineated target and organ at risk volumes and dosimetry | Up to 2 years
  Will be compared between the plans generated using the immediate post-op MRI versus (vs.) MR simulation. A Kolmogorov-Smirnov test will be used to assess distributional (histogram) changes between the two scenarios.
Cumulative dosimetric differences for the target volume and normal structures | Up to 2 years
  Cumulative dosimetric differences for the target volume and normal structures between an adaptive radiotherapy approach based on serial MR images vs. the conventionally delivered radiotherapy plan. A Kolmogorov-Smirnov test will be used to assess distributional (histogram) changes between the two scenarios.

SECONDARY OUTCOMES:
Incidence and temporal relationship of tumor progression between surgery and radiation therapy | Up to 2 years
  Specifically, the rate of change in volume between surgery and radiation therapy (RT) will be measured and reported.
Local tumor control | At 6 months post-treatment
  Local control is defined as stable disease, partial response or complete response using Response Assessment in Neuro-Oncology (RANO) criteria.
Local tumor control | At 12 months post-treatment
  Local control is defined as stable disease, partial response or complete response using RANO criteria.
Overall survival (OS) | From the date of start of radiation to the date of death, assessed up to 2 years
  A Cox proportional hazards regression model will be constructed to associate post-op progression with OS, after adjusting for age, IDH mutation, Karnofsky performance status and extent-of-resection.
Changes in co-registration accuracy under the two settings | Baseline up to 2 years
  A paired t-test (or a nonparametric analog) will be used to assess changes in co-registration accuracy under the two settings (post-op MRI vs. newly acquired MRI prior to radiation therapy).
Difference in reported pseudoprogression | Up to 6 weeks after completion of radiation
  Will determine the difference in the reported incidence of pseudoprogression at first follow-up after completion of 6 weeks of radiation when the immediate post-resection MRI is used as the baseline vs. newly acquired MRI prior to radiation therapy as the baseline. A binomial test of proportions between reported pseudo-progression in postsurgical MRI vs. baseline pre-radiation MRI with contrast will be performed.
Dosimetric differences | Up to 2 years
  Will be assessed via paired t-test (or a nonparametric analog).

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Chung, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org